CLINICAL TRIAL: NCT03459274
Title: Feasibility of an Immersive Virtual Reality Based Biofeedback Intervention for Outpatients in Rheumatology: An Observational Cohort Study
Brief Title: Feasibility of an Immersive Virtual Reality Based Biofeedback Intervention for Outpatients in Rheumatology
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: AppliedVR Inc. (Industry); Attune Health Research, Inc. (Industry)
Responsible Party: Principal Investigator, Swamy Venuturupalli, MD, FACR, Cedars-Sinai Medical Center
Other Study IDs: Pro00049211
Record Dates: First submitted 2018-02-23; First posted 2018-03-08 (Actual); Last update posted 2018-05-31 (Actual); Status verified 2018-05

CONDITIONS: Rheumatoid Arthritis; Systemic Lupus Erythematosus; Spondyloarthropathy; Vasculitis
MeSH Terms: conditions — Arthritis, Rheumatoid; Lupus Erythematosus, Systemic; Spondylarthropathies; Vasculitis | interventions — Biofeedback, Psychology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- VR-Biofeedback Feedback Sharers: These participants would express either interest or a lack of interest in trying biofeedback/virtual reality therapy. They will be instructed on how to use the virtual reality equipment and program. Then, they will have the option to participate in the biofeedback/virtual reality experience, if they choose to do so, before sharing their feedback.
  Interventions: Device: VR-Biofeedback

INTERVENTIONS:
Device: VR-Biofeedback — The intervention uses a smart phone with a virtual reality app; a headset that connects to the phone and has goggles that contribute to the 3 dimensional, interactive, and surrounding aspects of the experience; headphones through which subjects hear calming sounds and guiding voices from the experience; an attached microphone that allows subjects to monitor their breathing and interact with their environment through their breath; and a heart rate monitor whose realtime data on variability has an affect on the virtual environment. The virtual reality experience guides subjects through deep breathing exercises. Subjects will attempt to match a certain slow breathing rate, and pulse and breathing rate will cause non-stressful changes to the environment.
  Other Names: Applied Virtual Reality; Virtual Reality; Biofeedback

SUMMARY:
The purpose is to study the use of virtual reality (VR) and biofeedback in rheumatology clinics to help manage chronic pain in patients with rheumatologic diseases. The objective is to know the usefulness of VR/biofeedback-based therapy in the clinic.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with Rheumatoid arthritis, Systemic Lupus Erythematosus, Seronegative Spondyloarthropathy, Myositis, Psoriatic Arthritis, vasculitis or other autoimmune conditions.
* Patients must be on a stable regimen of medications.
* Patients should have pain, measured at the time of entry using a Visual Analog scale, of >5/10 at least 4 days in the last 30 days

Exclusion Criteria:

* Patients who are deemed by the study team to be unable to use the VR headset and follow instructions for any reason.
* Patients who have a history of vertigo and/or dizziness
* Patients with a history of seizure disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with Rheumatoid arthritis, SLE, Seronegative Spondyloarthropathy, Myositis, Psoriatic Arthritis, vasculitis or other autoimmune conditions. Patients must be on a stable regimen of medications. Patients should have pain, measured at the time of entry using a Visual Analog scale, of >5/10 at least 4 days in the last 30 days.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2018-03-16 (Actual); Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Self-reported benefit of virtual reality-biofeedback experience | Within 10 minutes immediately after virtual reality experience completion
  In interview, subjects are asked to describe their perception of the level of benefit of the Virtual Reality-Biofeedback experience

SECONDARY OUTCOMES:
Self-reported interest to try the virtual reality-biofeedback experience | Within 10 minutes immediately before virtual reality experience start
  Patients who are consented and fit inclusion criteria are asked, in interview, if they would be interested in trying the virtual reality experience and providing a rationale for their choice.

CONTACTS AND LOCATIONS:
Overall Officials: Swamy R Venuturupalli, MD, FACR, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Attune Health, Beverly Hills, California, United States